CLINICAL TRIAL: NCT05438069
Title: German Inclisiran Network: Retrospective Registry of Patients Being Treated With the siRNA Inclisiran in Germany
Acronym: GIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: Universitätsklinikum Leipzig (Other); Charite University, Berlin, Germany (Other); Technische Universität Dresden (Other); Deutsches Herzzentrum Muenchen (Other); University of Rostock (Other); Ruhr University of Bochum (Other); Universitätsmedizin Mannheim (Other); LMU Klinikum (Other)
Responsible Party: Principal Investigator, Oliver Weingärtner, Clinical Professor, Jena University Hospital
Other Study IDs: 2021-2429
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with elevated LDL-cholesterol (hypercholesterolemia): Application of si RNA Inclisiran to reduce serum LDL-cholesterol levels.

SUMMARY:
The German Inclisiran Network is a registry of patients with hypercholesterinemia on treatment with the siRNA inclisiran in Germany

DETAILED DESCRIPTION:
The aim of this retrospective, multi-center analysis is to use individual patient data to determine the extent of the variability in LDL-C reduction in response to inclisiran administration in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with elevated LDL-C levels (hypercholesterolemia) on stable lipid-lowering drugs for at least one month prior to the application of the siRNA Inclisiran
* patients 18 years and older

Exclusion Criteria:

- patients who do not qualify for treatment with the siRNA inclisiran according to the G-BA (Gemeinsamer Bundesausschuß) in Germany.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -patients with elevated LDL-C levels (hypercholesterolemia), who are treated with the siRNA Inclisiran
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
LDL-C change | 3 months, 6 months, 12 months, 24 months
  LDL-C change in mg/dL / mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Weingaertner, MD, Principal Investigator — Jena University Hospital
Locations (1):
- Jena University Hospital, Jena, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data that will be shared:
  Study protocol and individual participant data underlying the results reported in the project report or article, after deidentification. Documents will be available 3 months after publication for 3 years for researchers submitting a structured application, after approval by a committee. Data will be made available for all types of analyses that produce results in the approved application. Requests should be sent informally to oliver.weingaertner@med.uni-jena.de. A data agreement must be signed for access to the data.
Supporting Information: Study Protocol, SAP
Time Frame: 3 months after publication for 3 years
Access Criteria: Data that will be shared:
  Study protocol and individual participant data underlying the results reported in the project report or article, after deidentification. Documents will be available 3 months after publication for 3 years for researchers submitting a structured application, after approval by a committee. Data will be made available for all types of analyses that produce results in the approved application. Requests should be sent informally to oliver.weingaertner@med.uni-jena.de. A data agreement must be signed for access to the data.